CLINICAL TRIAL: NCT04842773
Title: MESSAge Study : Ultrasound Measurement of Sarcopenia in the Elder Subject
Brief Title: Ultrasound (US) Measurement of Sarcopenia in the Elder Subject
Acronym: MESSAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-AOI-09
Record Dates: First submitted 2021-04-07; First posted 2021-04-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- US measurement of sarcopenia (Experimental)
  Interventions: Diagnostic Test: Ultrasound measurement

INTERVENTIONS:
Diagnostic Test: Ultrasound measurement — Ultrasound measurement of sarcopenia in an elderly population

SUMMARY:
Sarcopenia is a generalized, progressive and multifactorial muscle impairment, causing multiple pathologies and their consequences such as falls, fractures, dependence, worsening of cognitive disorders and death. Interventions to combat the progression of sarcopenia should be introduced as soon as clinically suspected, based on functional tests to measure muscle strength. Diagnostic confirmation of sarcopenia can be done using several validated methods of estimating muscle mass: magnetic resonance imaging (MRI), computed tomography (CT), biphotonic absorptiometry (DEXA) or bio-impedanceometry. Their availability in clinical routine remains limited due to their high costs and/or lack of accessibility depending on the place of practice. On the other hand, there are certain pitfalls for carrying out these various examinations, in connection with several common clinical problems in the study population: mobility disorders and neurodegenerative disorders disabling for transport and access to the examination table for imaging examinations, hydration disorders distorting measures for bio-impedancetry.

Previous studies suggest that ultrasound may be as effective a tool as previous methods for diagnostic confirmation of sarcopenia. Because of its non-invasive and non-irradiating nature, its affordability, its short duration of realization, its availability and its low constraints of realization, the ultrasound could help to remove some of the current limits to the diagnostic confirmation of sarcopenia.

The investigators hypothesis is that ultrasound can be used to implement a simple and reliable protocol for assessing sarcopenia in the elderly. It could also be used to detect sarcopenia at an early stage ("presarcopenia") while the decrease in muscle mass is not yet accompanied by a decrease in skeletal muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 or older
* SARC-F > 4
* Decrease in muscle strength: grip strength <27 kg for men and <16 kg for women; and/or Chair stand test < 15 seconds
* Patient affiliated or beneficiary of a social security plan
* Patient who has signed informed consent beforehand

Exclusion Criteria:

* Neurocognitive disorder preventing the expression of informed consent
* Lack of a measurement site (muscle resection or amputation)
* Impossibility or contraindication to strict dorsal and/or ventral decubitus
* Any associated neuromuscular pathology that may alter muscle composition and trophicity
* Wearing a pacemaker
* Any state of water inflation or dehydration
* History of surgery on the studied lower limb less than 6 months old
* Patients protected by law under guardianship or under curate, or unable to participate in a clinical study under Article L. 1121-16 of the French Code of Public Health

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Combinaison of US measurements | 1 day
  To determine the most relevant combination of ultrasound measurements, the investigators will assess the muscles thickness in centimeters.

SECONDARY OUTCOMES:
Inter-operator reproductibility | 1 day
  To assess inter-operator reproducibility
Muscle elasticity | 1 day
  To explore whether muscle elasticity is a relevant ultrasound measure for assessing sarcopenia in an elderly geriatric population. Muscles elasticity will be assessed in meter/seconde.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, Provence-Alpes-Côte d'Azur Region, France

IPD SHARING:
Plan to Share IPD: No